CLINICAL TRIAL: NCT01043952
Title: Use of Bispectral Index (BIS) Monitoring of Anaesthesia With Propofol and Remifentanyl in Pediatric Patients in Ear Nose and Throat Surgery: Are There Clinical Advantages?
Brief Title: Use of Bispectral Index (BIS) for Monitoring of Total Intravenous Anaesthesia in Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment.
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Piergiorgio Bresil, MD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20090035
Record Dates: First submitted 2010-01-04; First posted 2010-01-07 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Anesthesia, General
Keywords: Propofol; Remifentanil; Bispectral Index Monitor
MeSH Terms: interventions — Propofol; Remifentanil; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients receive general anesthesia with Propofol and Remifentanil following clinical practice.
  Stratification by age (1-3 y, 4-11y, 12-17y, 18-65y) will be performed to ensure balanced allocation of age groups and allow for identification of age and weight specific effects.
  Stratification by operation type will be performed to ensure the identification of the effects of the duration of anaesthesia and of the use of longer acting opioids (Fentanyl) on outcome parameters.
  Interventions: Drug: Propofol; Drug: Remifentanil
- Bispectral Index Monitor (Experimental): Patients receive a general anesthesia with Propofol and Remifentanil where the amount of anesthetics administered is decided taking into consideration the Bispectral Index Monitor.
  Stratification by age (1-3 y, 4-11y, 12-17y, 18-65y) will be performed to ensure balanced allocation of age groups and allow for identification of age and weight specific effects.
  Stratification by operation type will be performed to ensure the identification of the effects of the duration of anaesthesia and of the use of longer acting opioids (Fentanyl) on outcome parameters.
  Interventions: Drug: Propofol; Drug: Remifentanil; Device: Bispectral Index Monitor

INTERVENTIONS:
Drug: Propofol — Propofol is used as an anesthetic drug on all patients, with the dosing depending on patient age, weight, body mass index, general status, the hemodynamic and neurophysiological response to the previously administered dose and the degree of surgical stimulation, and in the Bispectral Index Monitor arm, depending on the BIS values.
Drug: Remifentanil — Remifentanil is used as analgesic drug, as a part of the total intravenous anaesthesia, on all patients, with the dosing depending on patient age, weight, body mass index, general status, the hemodynamic and neurophysiological response to the previously administered dose and the degree of surgical stimulation, and in the Bispectral Index Monitor arm, depending on the BIS values.
  Other Names: Ultiva
Device: Bispectral Index Monitor — Bispectral Index Monitor (BIS monitor integrated in the IntelliVue Patient monitor MP70, Philips) is used to monitor the depth of anesthesia. The values this monitor reports are used as an aid in evaluating the response of the single patient to the administered anesthetics, and as a guide in adjusting the dosing of anesthetics. We follow the algorithm from: http://www.biseducation.com/assets.aspx?ac=1 (ASA Practice Advisory White Paper)
  Arms: Bispectral Index Monitor

SUMMARY:
The objective of the study is to determine wether the use of the Bispectral Index Monitor (BIS) as a method to guide anaesthesia for children in different groups of age, undergoing ear nose and throat surgery anaesthetized with an infusion of Propofol and Remifentanil with an high dose of Remifentanil (0,5-2 mcg/kg/min), can lead to a reduction in the time needed for extubation and in the amount of anesthetics used.

DETAILED DESCRIPTION:
The participants to the study are patients undergoing the following operations: Tonsillectomy, Adenoidectomy, Microlaryngoscopy, Bronchoscopy, Esophagoscopy, Myringoplasty, Myringotomy with positioning of a tube.

All these procedures are performed with the patient receiving a general anesthesia with and infusion of Propofol and Remifentanil. Muscle relaxants and inhaled anesthetics are not used.

The patients undergoing a Tonsillectomy will receive a supplementary opioid analgesic (Inj. Fentanyl iv, 3mcg/kg) at the end of the surgical procedure. Patients undergoing the other operations receive intraoperative Paracetamol and NSAID for postoperative pain treatment.

Stratification by age (1-3y, 4-11y, 12-17y, 18-65y) will be performed to ensure balanced allocation of age groups and allow for identification of age and weight specific effects. Stratification by operation type will be performed to ensure the identification of the effects of the duration of anaesthesia and of the use of longer acting opioids (Fentanyl) on outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 or 2
* General anesthesia for the following operations: Tonsillectomy, Adenoidectomy, Myringoplasty, Myringotomy with tube placement, microlaryngoscopy, bronchoscopy and esophagoscopy.

Exclusion Criteria:

* Psychiatric disorder
* Use of psychotherapeutic, antiepileptic, antiarrhythmic drugs
* Chronic use of opioids
* Intake of more than 21 alcoholic drinks/week
* Missing informed consent

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Time to extubation since the interruption in the administration of anaesthetics. | 30 minutes-3 hours

SECONDARY OUTCOMES:
Consumption of Remifentanil at induction and during maintenance of general anesthesia. | 30 minutes-3 hours
Average BIS during the surgical procedure | 30min-3hours
  Experimental arm: the anesthetist can read the values on the anaesthesia monitor and use them together with other clinical parameters to adjust the depth of the anaesthesia. Control arm: the BIS values are recorded in an hidden window of the anaesthesia monitor (they are not immediately available to the anesthetist), and are collected only at the end of the anaesthesia from a third person.
Consumption of Propofol during the induction and maintenance of anesthesia. | 30 minutes-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Piergiorgio Bresil, MD, Principal Investigator — Aalborg Hospital, 4th dept. of Anaesthesiology Region Nordjylland; Per H Lambert, MD, Study Director — Aalborg Hospital, 4th. dept. of Anaesthesiology Region Nordjylland
Locations (1):
- Aalborg Hospital, 4th. dept of Anaesthesiology, Division for Ear Nose and Troath anaesthesia, Aalborg, Nord Jylland, Denmark

REFERENCES:
- [Derived] Bresil P, Nielsson MS, Malver LP, Kraemer K, Schjorring O, Dethlefsen C, Lambert PH. Impact of bispectral index for monitoring propofol remifentanil anaesthesia. A randomised clinical trial. Acta Anaesthesiol Scand. 2013 Sep;57(8):978-87. doi: 10.1111/aas.12158. Epub 2013 Jul 15. PMID 23855759